CLINICAL TRIAL: NCT06051357
Title: An Multicenter, Randomized, Open-label Proof of Concept Study to Assess the Efficacy, Safety of HRS-5965 in Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: Proof of Concept Study to Assess the Efficacy, Safety of HRS-5965 in Patients With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-202
Record Dates: First submitted 2023-09-05; First posted 2023-09-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: HRS-5965 tablets
- Treatment group B (Experimental)
  Interventions: Drug: HRS-5965 tablets

INTERVENTIONS:
Drug: HRS-5965 tablets — HRS-5965 tablets for 12 weeks

SUMMARY:
This is a multicenter, randomized, open-label phase II clinical trial. A total of 24 patients with paroxysmal nocturnal hemoglobinuria naïve to complement inhibitor therapy were included. Subjects were treated with HRS-5965 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PNH confirmed by flow cytometry with clone size ≥ 10%.
2. Have not received complement inhibitor therapy ;
3. LDH > 1.5×ULN;
4. Hemoglobin level < 10 g/dL.

Exclusion Criteria:

1. Known or suspected hereditary or acquired complement deficiency;
2. Patients with laboratory evidence of bone marrow failure (reticulocytes <100x109/L; platelets <30x109/L; neutrophils <0.5x109/L);
3. Presence or suspicion of a systemic active bacterial, viral, or fungal infection (based on judgment of the investigator) within 2 weeks prior to the first dose of HRS-5965;
4. History of infection with capsular bacteria (e.g., meningococcus, pneumococcus, etc.)
5. Positive of HIV, HBsAg or HCVAb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin. | 12 weeks

SECONDARY OUTCOMES:
Changes in LDH. | 12 weeks
Changes in haptoglobin. | 12 weeks
Changes in bilirubin. | 12 weeks
Changes in reticulocyte counts. | 12weeks
Changes in C3 complement fragment deposition. | 12 week
Percentage of patients who did not receive a blood transfusion. | 12 weeks
Number of RBC units of transfused. | 12weeks
Incidence and severity of adverse events | 16 weeks
Incidence of thromboembolic events. | 16 weeks
Plasma concentration of HRS-5965. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Blood Disease Hospital of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided